CLINICAL TRIAL: NCT05703685
Title: [18F]PF-06445974 to Image PDE4B in Major Depressive Disorder Using PET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000676; 000676-M
Record Dates: First submitted 2023-01-27; First posted 2023-01-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12-04

CONDITIONS: Depression
Keywords: PET Imaging; Depression; Phosphodiesterase-4
MeSH Terms: conditions — Depression | interventions — apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- one arm (Other): All subjects will receive the same testsGroup D will have a baseline and block with apremilastGroup A & D will have a lung scan
  Interventions: Radiation: Lung scan; Drug: Apremilast; Drug: 18F-PF-06445974

INTERVENTIONS:
Radiation: Lung scan — Immediately after the brain scan
Drug: Apremilast — Oral administration of apremilast
Drug: 18F-PF-06445974 — Injected IV followed by PET scanning

SUMMARY:
Background:

Major depressive disorder (MDD) is a psychiatric condition. People with MDD have occasional bouts of depressive symptoms; these bouts are called major depressive episodes (MDEs). Researchers want to know if people having MDEs have lower levels of an enzyme called PDE4B in their brains.

Primary Objective: To determine whether PDE4B is reduced in the brains of individuals with MDD experiencing a major depressive episode (MDE). Secondary Objectives: To determine the optimal length of scanning and the retest variability and reliability of [18F]PF-06445974, and whether PDE4B binding correlates with clinical rating scales. To measure if PDE4B radioligand binding can be blocked by taking apremilast.

Eligibility:

People aged 18-70 years with MDD. Healthy volunteers are also needed.

Design:

Participants will have up to 5 clinic visits.

Participants will be screened. They will have a physical exam with blood tests. They will have a test of their heart function. Some participants may have a psychiatric assessment; they will answer questions about their state of mind and related topics.

Participants will have magnetic resonance imaging (MRI) of the brain. They will lie on a table that slides into a metal cylinder.

Participants will have a positron emission tomography (PET) scan. A needle will be used to guide a thin plastic tube (catheter) into a vein in one arm. An experimental substance called a radioactive tracer ([18F]PF-06445974) will be injected through the catheter. Participants will lie on a table that slides into a doughnut-shaped machine. The scan will last up to 4 hours with a 15-minute break.

Participants blood pressure, heart rate, and breathing will be monitored before, during, and after the PET scan. A second catheter will be inserted in the artery of the wrist so blood can be drawn during the scan.

Some participants may return for a second PET scan; have a lung scan or receive apremilast.

https://nimhcontent.nimh.nih.gov/start/surveys/?s=KE88DXXPLDFHHTF8

DETAILED DESCRIPTION:
Study Description:

This study will examine whether phosphodiesterase 4B (PDE4B) can be accurately quantified in the human brain and whether it is reduced in the brain of individuals with major depressive disorder (MDD).

Objectives:

Primary Objective:

To determine whether PDE4B is reduced in the brains of individuals with MDD experiencing a major depressive episode (MDE).

Secondary Objectives:

To determine the optimal length of scanning and the retest variability and reliability of [18F]PF-06445974, and whether PDE4B binding correlates with clinical rating scales.

Endpoints:

Primary Endpoint: measurement of PDE4B density (distribution volume VT) in the brains of individuals with MDD compared to healthy volunteers

Secondary endpoints:

1. To determine the optimal length for PDE4B scans with [18F]PF-06445974 PET scans in healthy volunteers
2. To measure whole-brain VT of PDE4B in a retest setting.
3. To assess the relationship between clinical rating scales and PDE4B binding.
4. To measure the blockade of PDE4B radioligand binding in brain after oral administration of apremilast.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients: In order to be eligible for this study, MDD participants must meet all of the following criteria:

* 18 to 70 years of age.
* Female participants of childbearing potential must be using a medically acceptable means of contraception.
* Be in good general health as evidenced by medical history and physical examination. Stable medical conditions as assessed by their primary care provider (PCP) and/or in-house clinician are permitted to join the study.
* Each participant must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
* All participants must have undergone a screening assessment under protocol 01-M-0254, The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Participants .
* Participants must fulfill DSM-5 criteria for major depression (MDD) without psychotic features, as based on clinical assessment and structured diagnostic interview (SCID-P).
* Participants must have an initial score on the MADRS >= 18 or HAM-D >= 15 within one week of study entry.
* Participants must be experiencing an MDE lasting at least four weeks.
* All MDD participants must have a PCP or psychiatrist in the community.
* Participants must have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Participants must agree to adhere to the lifestyle considerations.

Healthy Controls: In order to be eligible to participate in this study, control subjects must meet all of the following criteria:

* Aged 18 to 70 years old.
* Female participants of childbearing potential must be using a medically acceptable means of contraception.
* Able to provide informed consent.
* Be in good general health, as evidenced by medical history and physical examination, and have no cognitive impairment.
* Be enrolled in 01M0254, The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17M0181, Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies .
* Have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Participants with MDD who meet any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen). Any lab value that is two-times the upper limit or even lower values in the investigator s judgment. Creatinine level >1.3 mg/dL.
* Participants must be free of all prohibited medications for at least two weeks (5 weeks for aripiprazole, brexpiprazole, fluoxetine) prior to screen visit. These medications include antidepressants, antipsychotics, anxiolytics, psychotropic drugs not otherwise specified

(including herbal products), and sedatives/hypnotics.

* Current psychotic features, a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-5.
* Participants with a history of psychiatric inpatient hospitalization within the past year.
* Participants with a history of DSM-5 substance use disorder (except for caffeine or nicotine dependence) within the preceding three months. In addition, participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function of daily life.
* Participants who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
* Participants with suicidal ideation within the past 6 months.
* Participants with suicidal behavior within the past 12 months.
* Participants who have a history of aggressive behavior towards others.
* Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
* HIV infection.
* Pregnancy.
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
* Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

Healthy controls who meet any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).
* Participants must be free of all prohibited medications or at least two weeks (5 weeks for aripiprazole, brexpiprazole, fluoxetine) prior to screen visit. These medications include antidepressants, antipsychotics, anxiolytics, psychotropic drugs not otherwise specified (including herbal products), and sedatives/hypnotics.
* Participants with a history of DSM-5 substance use disorder (except for caffeine or nicotine dependence) within the preceding three months. In addition, participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function of daily life.
* Participants who have a history of major depressive disorder.
* Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
* HIV infection.
* Pregnancy.
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
* Use of cytochrome P450 enzyme inducers (e.g. rifampin, phenobarbital, carbamazepine, phenytoin).
* Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2028-10-03 (Estimated); Study Completion 2029-04-11 (Estimated)

PRIMARY OUTCOMES:
To measure distribution volume | 36 months
  Target quantification

SECONDARY OUTCOMES:
To determine the optimal length | 36 months
  Target quantification
To measure whole-brain distribution volume in retest | 36 months
  Target quantification
measure clinical rating scales and PDE4B binding | 36 months
  Assess the severity of depression

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be submitted to ClinicalTrials.gov and OpenNeuroPET with consent.
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000676-M.html